CLINICAL TRIAL: NCT03823521
Title: A Multi-Center, Open Label, Single Group, Observational Study to Investigate the Effects of Training on the Administration of Cardioplexol™
Brief Title: Observational Study to Investigate the Effects of Training on the Administration of Cardioplexol™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cardio Technologies AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCT-Cpx-004
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Bypass Surgery; Valve Surgery
Keywords: Cardioplegic Solutions
MeSH Terms: interventions — Cardioplegic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardioplexol™- Cardioplegia Solution (Experimental): Cardioplexol™ will be used as cardioplegic solution in cardiac surgery
  Interventions: Drug: Cardioplegia Solution

INTERVENTIONS:
Drug: Cardioplegia Solution — Cardioplexol™ will be adminstered in cardiac surgery as cardioplegic solution
  Other Names: Cardioplexol™

SUMMARY:
This is a multi-center, open label, single group, observational study designed to evaluate the effects of a Cardioplexol™ preparation and administration training program proposed to cardiac surgeons and cardiotechnicians inexperienced in the use of Cardioplexol™.

The training program aims at increasing the efficacy of Cardioplexol administration while reducing the risk of false manipulations. During the training possible risks and consequences of incorrect applications as well as the measures to take in case of administration error, are discussed. The training program includes one standardized theoretical part and one practical part consisting of a direct intra-operative coaching of surgeons practicing their first 2 operations.

The effect of the training will then be assessed by evaluating each trained surgeon's 4 next consecutive patients operated with Cardioplexol and without the coach.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 80 years of age;
* The patient's pre-operative evaluation indicates the need for a primary elective cardiac coronary artery bypass graft (CABG) operation and/or a cardiac valve repair/replacement;
* The operation can be carried out via a full sternotomy, under cardiac arrest and under the assistance of a heart lung machine;
* Patients who provide signed written informed consent.

Exclusion Criteria:

* Pre-operative EF of less than 30%;
* Pre-operative IABP;
* Pre-operative catecholamine support;
* History of myocardial infarction within less than 7 days;
* Previous history of cardiac surgery, including the implantation of a pace maker or an ICD;
* Active myocarditis and/or endocarditis;
* Aortic valve insufficiency severity grade more than 1;
* Under dialysis;
* Pre-operative serum creatinine value of more than 2.0 mg/dl;
* Known hematologic disorder;
* Treatment with anti-vitamin K;
* History of HIT;
* Participating in a concomitant research study of an investigational product;
* Pregnant or lactating;
* Intravenous drug user, alcohol abuser, prisoner, institutionalized, or is unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Major Deviation in Cardioplexol application | During surgery
  Number of major deviations from the application of Cardioplexol™ as determined by the pre-specified training documentation (incorrect volume of initial dose, incorrect volume of second/third/fourth dose, incorrect duration of injection of initial dose, incorrect timing of application of initial dose, incorrect timing of application of second/third/fourth dose).

SECONDARY OUTCOMES:
TnT Values | During the first 24 hours following myocardial reperfusion
  Development of concentration of blood Troponin T values measured by the local hospital laboratory
CK-MB Values | During the first 24 hours following myocardial reperfusion
  Development of concentration of blood Creatin Kinase - isoenzyme MB (muscle-brain) values measured by the local hospital laboratory
Complete Cardiac Arrest | During Surgery
  Time between the aortic cross-clamping and the complete cardiac arrest
Catecholamine | During during aortic cross-clamping and during the first 24 hours
  Cumulative dose of catecholamines
Defibrillation rate | During surgery
  Defibrillation rate after aorta unclamping and coronary reperfusion.
ICU stay | During follow-up phase after surgery up to 35 days
  Duration of ICU stay
Mortality | During the first 24 hours following coronary reperfusion
  Number of patients, who died

CONTACTS AND LOCATIONS:
Locations (6):
- Austria (4):
  - Universitätsklinik Innsbruck, Innsbruck
  - Universitaetsklinikum Salzburg, Salzburg
  - Universitaetsklnikum St. Pölten, Sankt Pölten
  - Krankenhaus Hietzing, Vienna
- Germany (2):
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitaetsklinikum Frankfurt, Frankfurt

REFERENCES:
- [Derived] Tevaearai Stahel HT, Taheri N, Winkler A, Hohlfeld J, Dietl W, Starck C, Van Linden A, Bidovec J, Imhof A, Carrel TP, Voet B, Walther T, Seitelberger R, Grimm M, Holzinger C, Grabenwoger M. A multi-center, open label, single group, observational clinical trial to investigate the effects of training on the administration of Cardioplexol. Front Cardiovasc Med. 2025 May 26;12:1588088. doi: 10.3389/fcvm.2025.1588088. eCollection 2025. PMID 40491721